CLINICAL TRIAL: NCT05096858
Title: Assessment of the Effect of Continuous Glucose Monitorization on Glycemic Variability and Insulin's Prescription in Hospitalized Patients With COVID-19
Brief Title: Continuous Glucose Monitorization in Hospitalized Patients With COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Sponsor
Other Study IDs: 3066
Record Dates: First submitted 2021-09-13; First posted 2021-10-27 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2023-09

CONDITIONS: Diabetes Mellitus; Covid19
MeSH Terms: conditions — Diabetes Mellitus; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
DM2 is a major comorbidity of COVID-19. It has been observed that subjects with DM2 require more medical interventions, have a significantly higher mortality (7.8% versus 2.7%) and injuries of multiple organs that the individuals not diabetics.

In situations of glycemic variability, phenomena of oxidative stress and activation of protein kinase C can be initiated , through the release of pro-inflammatory cytosines , which could induce microvascular damage .Patients with diabetes and COVID-19 were shown to be more likely to develop serious or critical illness with more complications, and to have higher incidence rates of antibiotic therapy, non-invasive and invasive mechanical ventilation, and death (11.1% vs. 4.1%).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed COVID-19 pneumonia
* Diabetes mellitus

Exclusion Criteria:

* Less than 3 days of hospital care

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults living with diabetes and suffering from COVID19 pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Glucose variability | For up to two weeks, during hospitalization
  Percentage of time within the ADA recommended range
Insulin use | For up two weeks, during hospitalization
  Average daily UI of insulin per patient

CONTACTS AND LOCATIONS:
Overall Officials: ALFONSO GULIAS HERRERO, Principal Investigator — INCMNSZ
Locations (1):
- National Institute of Medical Sciences and Nutrition Salvador Zubiran, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided